CLINICAL TRIAL: NCT05157256
Title: Monitoring of Anti-SARS-CoV-2 (COVID 19) and Encapsulated Vaccination in a Cohort of Patients With Thalassemic and Falcemic Syndromes
Brief Title: Monitoring of Anti-SARS-CoV-2 (COVID 19) and Encapsulated Vaccination Patients With Thalassemic and Falcemic Syndromes
Acronym: HEMOGLOB-VAX
Status: Active, not recruiting | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_HEMOGLOB-VAX_COVID19
Record Dates: First submitted 2021-12-10; First posted 2021-12-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2 Infection, Thalasemmie, SCD
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is an urgent need to rapidly evaluate anti-Covid 19 vaccination treatments, in terms of immune response (humoral and cell-mediated) together with the verification of the effectiveness of the vaccine in preventing SARS-CoV-2 infection in thalassemic subjects.

It is also necessary to increase scientific knowledge in order to improve clinical practice to have presence responses and maintenance extent of the response to vaccinations against encapsulated bacteria carried out previously.

The objectives of the main study are:

1. Evaluate the appearance, extent, and duration of humoral response (antibodies) to the anti-SARS-CoV-2 vaccine;
2. Assess the incidence of positive cases after vaccination.

The objective of the first sub-study is:

- Evaluate the appearance, extent, and duration of cellular response (T lymphocytes and B lymphocytes) to the anti-SARS-CoV-2 vaccine based on age groups and the presence/absence of hypo/asplenia.

The objective of the second sub-study is:

- Evaluate the presence and extent of the response to previous vaccinations to encapsulated bacteria.

DETAILED DESCRIPTION:
This is a non-profit multicenter observational study, coordinated by the Department of OncoHematology,Cell Therapy, Gene Therapies and Hematopoietic Transplantation of the Bambino Gesù Children'sHospital, IRCCS which provides for the collectionof clinical data of patients with an established diagnosis of TDT and SCD after the administration of the anti-SARS-CoV-2vaccine.

As this is a prospective study for medium-term assessments, it is expected to last no less than 18 months. The duration of the prospective observation will start from April 2021 for the duration of 12 months.

Setting

The following will be enrolled:

* for the main study patients diagnosed with TDT and SCD even if they have previously contracted SARS-CoV-2 infection;
* for the first substudy, patients with TDT and SCD diagnosis will be enrolled, divided by presence/absence of hypo/asplenia;
* for the second substudy, patients diagnosed with TDT and hypo/asplenic SCD will be enrolled.

The Scientific Committee of the project discussed and approved a dataset that will be collected by local centers, the pseudo-anonymized data of patients collected in a special e-CRF.

The participating centers are:

- Rome, Brindisi, Cagliari, Genoa, Ferrara, Milan, Naples, Palermo Turin, Verona.

The Italian Society of Thalassemia and Hemoglobinopathies (SITE) in its role as a scientific society of reference for the pathology will act as Promoter of the experimentation and the ForAnemia Foundation, a non-profit organization, is also identified as a funder of the present study.

The project will be developed through the creation and validation of a data collection card in which the clinical data relating to all patients with the characteristics of inclusion in the participating centers will be entered.

The data to be entered include characteristics of the patient, in addition to epidemiological data (sex, age) and clinical data (diagnosis), pre-existing comorbidities, indication of iron overload, drugs administered. Data analysis will be primarily descriptive.

It is accepted in advance that this protocol may require repeated modifications to conform to the evolution of knowledge about the pandemic, the complication rate and the therapeutic scenario. A high degree of adaptation is therefore expected, which will be rigorously discussed with the independent data monitoring committee that will be appointed immediately after the approval of the protocol.

Study population Patients with TDT and SCD. Inclusion criteria

Main study and first substudy:

* Patients with advancedTDT and SCD diagnosis, age > 18 years
* signature of informed consent.

Second substudy:

* Splenectomized patients withTDT and SCD diagnosed, age > 18 years
* signature of informed consent. Exclusion criteria No signature informed consent. Results of the Study

The following variables will be measured:

* anti_N Antibody Value
* Anti-RBD values
* memory andi-trimeric Spike IgG in total memory (% of total IgG memory)
* Immunity value T (IFN-g) Variables Samples for the analysis of humoral and cell-mediated response will be collected before vaccination (T0), at booster (T1), between 14 and 21 days after recall (T2) and after 12, 24 and 52 weeks after vaccination.

Sampling before vaccination (T0) can be collected up to 5 days before vaccination. Sampling prior to administration of the booster (T1) may be collected up to 5 days in advance.

Withdrawals at weeks 12, 24, 52 will be performed with a tolerance of 10 days.

- The analysis of the presence of specific antibodies (IgG) to N and S viral antigens will be carried out by CMIA method. The analysis of both antibodies will allow to evaluate the response to the vaccine (anti-S antibodies) and a possible natural exposure/infection (anti-N antibodies). In patients who present anti-S antibodies, neutralizing titiness measurement will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

Main study and first substudy:

* Patients with advancedTDT and SCD diagnosis, age > 18 years
* signature of informed consent.

Second substudy:

* Splenectomized patients withTDT and SCD diagnosed, age > 18 years
* signature of informed consent.

Exclusion Criteria:

No signature informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with TDT and SCD.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the appearance, extent, and duration of humoral response (antibodies) to the anti-SARS-CoV-2 vaccine; | through study completion, an average of 1 year
Assess the incidence of positive cases after vaccination. | through study completion, an average of 1 year
- Evaluate the appearance, extent and duration of cellular response (T lymphocytes and B lymphocytes) to the anti-SARS-CoV-2 vaccine based on age groups and the presence/absence of hypo/asplenia | through study completion, an average of 1 year
Evaluate the presence and extent of the response to previous vaccinations to encapsulated bacteria. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Azienda Ospedaliero-Universitaria S. Luigi Gonzaga, Orbassano, Torino, Italia, Torino, TO
  - Azienda Ospedaliera Universitaria Di Cagliari, Cagliari
  - Day Hospital della Talassemia e delle Emoglobinopatie - A.O.U. di Ferrara - Nuovo Ospedale S.Anna - Sede di Cona, Ferrara
  - Ospedali Galliera - S.S.D. Microcitemia, anemie congenite e dismetabolismo del ferro, Genova
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - Department of Women, Children and General and Specialist Surgery AOU-- University of Campania "Luigi Vanvitelli, Napoli
  - U.O.C. di Ematologia e Malattie Rare del Sangue e degli Organi Ematopoietici - Azienda Ospedaliera Ospedali Riuniti "Villa Sofia-Cervello" - Presidio Cervello, Palermo
  - Dipartimento OncoEmatologia, Terapia Cellulare, Terapie Geniche e Trapianto Emopoietico, Roma
  - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: Undecided